CLINICAL TRIAL: NCT07075952
Title: Testing FoodTraining (FoodT): A Mobile App to Train Inhibitory Control Towards Food and Augment Standard Treatment for People With Eating and Weight Disorders
Brief Title: Training App for Inhibitory Control Towards Food
Acronym: FoodT-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Principal Investigator, CARDI VALENTINA, Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AOP3416
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-07

CONDITIONS: Obesity &Amp; Overweight; Bulimia Nervosa; Binge-Eating Disorder
Keywords: App; Training; Inhibitory control; Bulimia Nervosa; Binge-Eating Disorder; Obesity
MeSH Terms: conditions — Obesity; Overweight; Bulimia Nervosa; Binge-Eating Disorder; Alzheimer Disease | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: This study will use a randomised controlled design to test the impact of food-specific inhibitory control training offered in addition to treatment as usual on eating behaviour, eating attitudes and several areas of individual functioning in people with bulimia nervosa, binge eating disorder or obesity.
Who Masked: Outcomes Assessor
Masking Description: Each participant will be assigned an identification code (ID-code) randomly generated by a computer. The outcome assessors will be blind to whether participants will be assigned to the experimental or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Condition (TAU + FoodTraining) (Experimental): Participants in the experimental condition will be asked to perform a food-specific inhibitory control training delivered through the FoodTraining App once a day for the first week and three times a week for the remaining three weeks, for five minutes each time.
  Interventions: Behavioral: Food-specific inhibitory control training delivered through the FoodTraining App
- Control condition (Active Comparator): Participants in the control group will be offered access to the FoodTraining App at the end of the 8-week follow-up.
  Interventions: Behavioral: Waiting list

INTERVENTIONS:
Behavioral: Food-specific inhibitory control training delivered through the FoodTraining App — Participants will complete one training session per day for the first week and three sessions per week for the following three weeks (4 weeks in total). Each session lasts about 5 minutes and includes 3 blocks of stimuli presentation. In each block, 32 images (8 low-energy-dense foods, 8 high-energy-dense foods, 16 neutral objects) are presented for 1500ms with a 500ms interstimulus interval. One-hundred ms after the image presentation, a red or green circle appears. Participants will have to tap the image when a green circle appears ("go" trials) and inhibit a response when a red circle appears ("no-go" trials). Low-energy-dense foods are always paired with "go" trials, high-energy-dense foods with "no-go" trials, and neutral objects with either "go" or "no-go" trials. After each block, participants receive feedback on mean accuracy and reaction time. Participants can personalise the training by selecting up to three categories of high-energy-dense foods to include.
  Arms: Experimental Condition (TAU + FoodTraining)
Behavioral: Waiting list — Participants allocated to the control condition will not have access to the FoodTraining App during the active phase of the study (8 weeks), but will be offered the opportunity to access the app at the end of the 8-week follow-up period. This ensures that all participants, regardless of group allocation, will have the chance to benefit from the intervention once data collection is complete.
  Arms: Control condition

SUMMARY:
The aim of this project is to test the feasibility, acceptability and clinical impact of a mobile app-based intervention (FoodTraining) to strengthen food-related inhibitory control over 4 weeks, in a sample of people with eating or weight disorders (i.e. obesity, binge-eating disorder (BED), or bulimia nervosa (BN)) receiving standard outpatient treatment (i.e., treatment as usual (TAU) encompassing guided self-help or psychotherapy, pharmacological therapy or diet). The training will be offered in addition to TAU (experimental group) and compared to TAU alone (control group).

Participants will complete questionnaires to measure eating behaviour, eating disorder psychopathology, symptoms of anxiety, depression and stress, social functioning and quality of life at baseline, 4 and 8 weeks. They will also complete momentary assessments using a mobile application (FoodTracker) to report on food intake along with related thoughts, emotions, and behaviours and will wear small, non-invasive sensors to track real-time fluctuations in glucose levels for 15 days.

Participants will also perform a food-related go-no go task and a food-related temporal discounting task at baseline, 4 and 8 weeks.

Finally, this study will pilot the use of a semi-structured interview to characterise the history of weight, the appetite system, eating-related habits in the family and learning of eating behaviours and attitudes in people with eating or weight disorders.

DETAILED DESCRIPTION:
The study aims:

* To establish the feasibility, acceptability and clinical impact of a food-specific inhibitory control training delivered through a mobile App (i.e., FoodTraining) over 4 weeks in a sample of patients with obesity, bulimia nervosa or binge-eating disorder (N = 113) offered in addition to TAU, compared to TAU alone;
* To test the acceptability and adherence to the ecological momentary assessments collected through the Food Tracker App and the sensors for glucose monitoring;
* To characterise history of weight, appetite system, eating-related habits in the family and learning of eating behaviours and attitudes in people with obesity presenting for weight loss treatment.

An a-priori power analysis performed on the G*Power software, indicated that 93 participants would be needed to detect a significant 2 (group) x 3 (time) within-between interaction effect on the primary outcome measure (emotional eating and uncontrolled eating) with a small to medium effect size (Cohen's f = 0.15), a statistical power of 1-β = .80, and at a significant level α = .05, assuming a correlation among repeated measures of r = .5. To account for possible drop-out, the number will be exceeded by 20%. The final sample size that will be recruited is 113 participants.

Patients will be recruited and assessed at baseline, 4 and 8 weeks follow-up from the University Hospital in Padova (i.e., Eating Disorders Unit and Obesity Management Unit).

Assessment phase

After providing written informed consent, participants will complete a questionnaire to collect demographic information, such as gender and age. Their weight and height will be measured by a clinician. Clinical information, such as diagnosis, psychiatric/medical comorbidities and ongoing treatment will be retrieved from hospital clinical records. Participants will complete the following self-report questionnaires, measures and computerised tasks:

* The Three Factors Eating Questionnaire (TFEQ): a 51-item self-report questionnaire to assess eating-related feelings and behaviours. It comprises three subscales: cognitive restraint (i.e., efforts and worries to regulate food intake to control body weight and shape), uncontrolled eating (i.e., tendency to lose control and overeat), and emotional eating (i.e., tendency to eat in response to emotional urges, both positive and negative);
* The Dutch Eating Behavior Questionnaire (DEBQ): a 33-item self-report questionnaire grouped in 3 subscales: emotional eating (i.e., eating in response to internal emotional factors like fear, anxiety and anger), external eating (eating in response to external stimuli such as the sight and smell of food) and restrained eating (eating less than desired to lose or maintain a particular body weight);
* The Food Cravings Questionnaire-Trait (FCQ-T): a validated self-report instrument designed to assess the frequency and intensity of food cravings as a stable individual characteristic. Comprising 39 items, the FCQ-T evaluates multiple dimensions of trait food craving, including emotional triggers, cognitive preoccupation with food, lack of control, and anticipation of positive reinforcement from eating. Higher scores indicate a greater tendency to experience food cravings;
* Eating Disorder Examination Questionnaire (EDE-Q): a 28-item self-report questionnaire designed to assess the range, frequency and severity of eating disorder features. It includes the following subscales: Restraint (i.e. dietary restriction and attempts to control food intake), Eating Concern (i.e. preoccupation with food, eating, and guilt related to eating), Shape Concern (i.e. dissatisfaction, overvaluation, and preoccupation with body shape) and Weight Concern (i.e. preoccupation with weight, desire to lose weight, and fear of weight gain) and an overall Global score;
* Binge Eating Scale (BES): a self-report questionnaire to assess the severity of binge eating behavior. It includes 16 items that measure both behavioral manifestations (e.g., loss of control during eating episodes) and emotional and cognitive aspects (e.g., feelings of guilt or distress related to overeating);
* Depression Anxiety Stress Scales, Short Version (DASS-21): a 21-items screening tool to assess symptoms of depression, anxiety, and stress. It comprises three subscales: (1) Depression subscale measuring hopelessness, low self-esteem, and low positive affect; (2) Anxiety subscale assessing autonomic arousal, musculo-skeletal symptoms, situational anxiety and subjective experience of anxious arousal; and (3) Stress subscale evaluating tension, agitation, and negative affect;
* Work and Social Adjustment Scale (WSAS): a 5-item questionnaire assessing the impact of a person's mental health difficulties on their ability to function in terms of work, home management, social leisure, private leisure and personal or family relationships;
* Food-related liking and wanting, emotional states, and urge to eat visual analogue scales (0-100) will be used for subjective ratings of liking, wanting, emotional states and urge to eat following food pictures presentation;
* Yale Food Addiction Scale (YFAS): a 25-item self-report questionnaire assessing food addiction levels (compulsive consumption of palatable and hyperpalatable food items, often high in sugar, fat and salt contents, with marked activation of the reward system, and clinically significant impairment or distress on several areas of functioning);
* Barratt Impulsiveness Scale-11 (BIS-11): a 30-item self-report questionnaire to measure trait impulsivity. It encompasses three main domains: attention impulsivity (i.e. cognitive instability and inability to focus), motor impulsivity (i.e. acting without thinking), and non-planning impulsivity (i.e. lack of future orientation or forethought);
* Computerised food-related go/no-go task: it is a widely used paradigm to assess food-related response inhibition. The task will be divided into 10 blocks. In half of the blocks the pleasant stimuli (no-go stimuli) will be images of palatable foods, while in the other 5 blocks, no-go stimuli will be images of animals. In all blocks, go-stimuli will be pictures of neutral objects (e.g. office supplies, furniture). Participants will be instructed to press the spacebar on the computer keyboard as quickly as possible when they see a go stimulus (object), and to refrain from pressing any key when they see a no-go stimulus (food or animals). Each block will include 20 trials for a total of 200 trials. Numbers of errors will be used to assess inhibitory control;
* Computerised food-related temporal discounting tasks (TD task): a computerized temporal discounting task involving food and money rewards. Participants will be asked to select their preferred food by choosing one of four alternatives, which will be presented during the tasks. After selecting the preferred rewards, they will complete two tasks in a counterbalanced order. In each trial, they will have to choose between a smaller immediate reward or a larger reward delayed by one of six time intervals: 2 days, 2 weeks, 1 month, 3 months, 6 months, or 1 year. Each delay block will consist of five choices, with the delayed reward fixed at 40 units and the immediate reward adjusted based on previous choices using a titration method. The order of the delay blocks will be randomized across participants. Participants will be instructed to imagine receiving the rewards at the specified times and told there are no right or wrong answers. The trials will start with an immediate reward of 20 units; if the immediate option is chosen, its amount decreases in the following trial, and if the delayed option is chosen, the immediate amount increases. The size of adjustments halves after each choice, refining the estimate of the immediate reward equivalent to the delayed reward. The final data from each TD task will be fitted to a hyperbolic discounting function, yielding a discount rate (k) that reflects the degree to which participants prefer immediate over delayed rewards (i.e. the higher the k, the stronger the preference for immediate rewards);
* A semi-structured interview developed by the research team will be used at baseline to characterise the history of weight, the appetite system, eating-related habits in the family and learning of eating behaviours and attitudes.

A mobile App (i.e. FoodTracker), will be used to track food consumption, eating behaviours and their emotional and cognitive correlates for 3 days. Participants will be asked to complete the EMAs before and after each meal, and will also be prompted to respond to the survey questions at three random time points during the day. As a measure of physiological correlates of food consumption, glycemic responses will be monitored over a 15-day period using the FreeStyle Libre 3 device (https://www.freestyle.abbott/it-it/products/freestyle-libre-3.html), for continuous glucose monitoring (CGM). This tool collects real-time data on physiological changes in glucose regulation by measuring interstitial glucose levels every minute via a small sensor worn on the back of the upper arm. The sensor captures fluctuations in glucose throughout the day and night, providing detailed information on glycemic variability, postprandial responses, and potential episodes of hypo- or hyperglycemia.

All participants will be assessed through online self-report questionnaires at the end of the intervention (week 4) and follow-up (week 8). At all time points, weight will be measured. At 4- and 8-week follow-up, participants will complete a subset of the measures completed at baseline: Dutch Eating Behavior Questionnaire (DEBQ); Three Factors Eating Questionnaire (TFEQ); Food Cravings Questionnaire-Trait (FCQ-T); Eating Disorder Examination Questionnaire (EDE-Q); Binge Eating Scale (BES); Depression Anxiety Stress Scales Short Version (DASS-21); Work and Social Adjustment Scale (WSAS); Food liking and wanting; Food-related go/no-go task; Food-related temporal discounting task.

Intervention phase

Participants will be randomly assigned to either:

• The experimental condition (TAU + food-specific inhibitory training) or the control condition (TAU only).

All participants will be instructed to download the Food Tracker app and complete the EMAs for three days after the baseline assessment and three days after the 4-week assessment.

Participants assigned to the TAU+FoodTraining group will have access to the FoodTraning App following the baseline EMAs. They will be asked to complete a session once a day for the first week and three times a week for the remaining three weeks.

Participants in the control group will be offered access to the FoodTraining App at the end of the 8-week follow-up.

Access to the FoodTraining and FoodTracker Apps will be free of charge for participants.

ELIGIBILITY:
Inclusion Criteria:

* BMI in the obesity range (>30) or a clinician-formulated diagnosis of binge eating disorder or bulimia nervosa;
* knowledge of Italian or English;
* access to a mobile device (e.g. smartphone, tablet).

Exclusion Criteria:

* visual impairment not corrected by glasses
* a diagnosis of psychosis;
* intellectual disability.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Between-group differences (experimental vs. control group) in changes in tendency to eat in response to emotional eating | baseline; 4-, and 8- week follow-up
  Emotional eating subscale of the Dutch Eating Behavior Questionnaire (DEBQ). Higher scores indicate a greater tendency to eat in response to internal emotional factors. Sum and mean of the scores for each subscale item: 1-2 = low level of that eating behaviour; 3 = medium level; 4-5 = high level.
Between-group differences (experimental vs. control group) in changes in uncontrolled eating behaviours | baseline; 4-, and 8- weeks follow-up
  Uncontrolled Eating subscale of the Three-Factor Eating Questionnaire (TFEQ). Higher scores indicate greater levels of the behaviour (Cognitive Restraint = 0-21; Uncontrolled Eating = 0-16; Emotional Eating = 0-14).

SECONDARY OUTCOMES:
Between-group differences (experimental vs. control group) in changes in eating disorder psychopathology | baseline; 4-, and 8- weeks follow-up
  Eating Disorder Examination Questionnaire (EDE-Q; total score. min=0; max=6, cut-off 4). Higher scores indicating increased eating difficulties.
Between-group differences (experimental vs. control group) in changes in frequency and severity of binge eating episodes | baseline; 4-, and 8- week follow-up
  Binge Eating Scale (BES), score range 0-46 (18-26= moderate bingeing; >/= 27= severe bingeing).
Between-group differences (experimental vs. control group) in liking of high calorie dense foods | baseline; 4-, and 8- weeks follow-up
  Visual analogue scale to rate the degree of food liking in response to images of unhealthy and healthy foods developed by the research team (score range 0-100).
Between-group differences (experimental vs. control group) in wanting of high calorie dense foods | baseline; 4-, and 8- weeks follow-up
  Visual analogue scale to rate the degree of food wanting in response to images of unhealthy and healthy foods developed by the research team (score range 0-100).
Between-group differences (experimental vs. control group) in urge to eat high calorie dense foods | baseline; 4-, and 8- weeks follow-up
  Visual analogue scale to rate the urge to eat in response to images of unhealthy and healthy foods developed by the research team (score range 0-100).
Between-group differences (experimental vs. control group) in food-related inhibitory control level | baseline; 4-, and 8- weeks follow-up
  Number of errors to the food-related go/no-go task.
Between-group differences (experimental vs. control group) in changes in preference for immediate food rewards as compared to money | baseline; 4-, and 8- weeks follow-up
  Hyperbolic discount-rate for food rewards as compared to money to the temporal discounting task.
Between-group differences (experimental vs. control group) in changes in food craving | baseline; 4-, and 8- weeks follow-up
  Food Cravings Questionnaire-Trait (FCQ-T), higher scores indicate higher difficulties.
Between-group differences (experimental vs. control group) in food-related unpleasant emotions | 3-day evaluation at baseline, repeated at 4-, and 8- weeks follow-up
  Longitudinal comparison of responses to EMAs (visual analogue scales developed by the research team 0-5).
Acceptability and adherence of the EMA assessments (FoodTracker) | 8- weeks follow-up
  At least average 70% of participants providing a score of 7 or higher on a 1-10 Likert scale measuring the perceived acceptability of the daily assessments.
Acceptability and adherence to glucose monitoring assessments | 8- weeks follow-up
  At least average 70% of participants providing a score of 7 or higher on a 1-10 Likert scale measuring the perceived acceptability of the daily assessments.
Impact of food addiction on the degree of changes in response to internal emotional factors in the experimental and control groups | baseline
  Emotional Eating subscale of the Dutch Eating Behavior Questionnaire (DEBQ). Higher scores indicate a greater tendency to eat in response to internal emotional factors. Sum and mean of the scores for each subscale item: 1-2 = low level of that eating behaviour; 3 = medium level; 4-5 = high level.
Impact of food addiction on the degree of changes in uncontrolled eating in the experimental and control groups | baseline
  Uncontrolled Eating subscale of the Three-Factor Eating Questionnaire (TFEQ). Higher scores indicate greater levels of the behaviour (Uncontrolled Eating = 0-16).
Impact of impulsivity on the degree of changes in eating in response to internal emotional factors in the experimental and control groups | baseline
  Emotional eating subscale of the Dutch Eating Behavior Questionnaire (DEBQ). Higher scores indicate a greater tendency to eat in response to internal emotional factors. Sum and mean of the scores for each subscale item: 1-2 = low levels; 3 = medium levels; 4-5 = high levels.
Impact of impulsivity on the degree of changes in uncontrolled eating in the experimental and control groups | baseline
  Uncontrolled Eating subscale of the Three-Factor Eating Questionnaire (TFEQ). Higher scores indicate greater levels of the behaviour (Uncontrolled Eating = 0-16).
Between-group differences (experimental vs. control group) in changes in anxiety, stress and depression symptoms | baseline; 4-, and 8- weeks follow-up
  The Depression Anxiety Stress Scales-21 (DASS-21): 3 subscales. Stress subscale: Normal: 0-10; Mild: 11-18; Moderate: 19-26; Severe: 27-34; Extremely severe: 35-42. Anxiety: Normal : 0-6, Mild : 7-9, Moderate:10-14, Severe: 15-19, Extremely severe: 20-42. Depression: Normal: 0-9, Mild : 10-12, Moderate : 13-20, Severe : 21-27, Extremely severe: 28-42.
Between-group differences (experimental vs. control group) in changes in social adjustment levels | baseline; 4-, and 8- weeks follow-up
  Work and Social Adjustment Scale (WSAS). Total score ranges from 0 to 40 (Scores >/= 20 indicates moderately severe or worse impairment. Scores between 10 and 20 are associated with significant functional impairment but less severe clinical symptomatology)
Adherence to the intervention (FoodTraining) | 4 weeks follow-up
  Number of times participants complete the training task (FoodTraining) throughout the 4-week period.
Feasibility of the intervention (FoodTraining) | 8- weeks follow-up
  At least 60% of participants completing a minimum of 70% of the training sessions.
Acceptability of the intervention (FoodTraining) | 8- weeks follow-up
  At least 80% of participants providing a score of 7 or higher on a 1-10 Likert scale measuring the perceived acceptability and usefulness of the training.

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Cardi, PhD, Principal Investigator — Department of General Psychology, University of Padova, Padova, Italy
Locations (1):
- Psychiatry Unit, University Hospital, Padova and Bariatric Unit, University Hospital, Padova, Padua, Padova, Italy

IPD SHARING:
Plan to Share IPD: No
A plan will be established by the research team for data sharing following publication of the first manuscript

REFERENCES:
- [Background] Dakanalis A, Zanetti MA, Clerici M, Madeddu F, Riva G, Caccialanza R. Italian version of the Dutch Eating Behavior Questionnaire. Psychometric proprieties and measurement invariance across sex, BMI-status and age. Appetite. 2013 Dec;71:187-95. doi: 10.1016/j.appet.2013.08.010. Epub 2013 Aug 30. PMID 23994503
- [Background] Schiff S, Amodio P, Testa G, Nardi M, Montagnese S, Caregaro L, di Pellegrino G, Sellitto M. Impulsivity toward food reward is related to BMI: Evidence from intertemporal choice in obese and normal-weight individuals. Brain Cogn. 2016 Dec;110:112-119. doi: 10.1016/j.bandc.2015.10.001. Epub 2015 Oct 30. PMID 26525096
- [Background] Presseller EK, Parker MN, Zhang F, Manasse S, Juarascio AS. Continuous glucose monitoring as an objective measure of meal consumption in individuals with binge-spectrum eating disorders: A proof-of-concept study. Eur Eat Disord Rev. 2024 Jul;32(4):828-837. doi: 10.1002/erv.3094. Epub 2024 Apr 3. PMID 38568882
- [Background] Rania M, Caroleo M, Carbone EA, Ricchio M, Pelle MC, Zaffina I, Condoleo F, de Filippis R, Aloi M, De Fazio P, Arturi F, Segura-Garcia C. Reactive hypoglycemia in binge eating disorder, food addiction, and the comorbid phenotype: unravelling the metabolic drive to disordered eating behaviours. J Eat Disord. 2023 Sep 19;11(1):162. doi: 10.1186/s40337-023-00891-z. PMID 37726785
- [Background] Cornier MA. A review of current guidelines for the treatment of obesity. Am J Manag Care. 2022 Dec;28(15 Suppl):S288-S296. doi: 10.37765/ajmc.2022.89292. PMID 36525676
- [Background] Carbine KA, Muir AM, Allen WD, LeCheminant JD, Baldwin SA, Jensen CD, Kirwan CB, Larson MJ. Does inhibitory control training reduce weight and caloric intake in adults with overweight and obesity? A pre-registered, randomized controlled event-related potential (ERP) study. Behav Res Ther. 2021 Jan;136:103784. doi: 10.1016/j.brat.2020.103784. Epub 2020 Dec 8. PMID 33316579
- [Background] de Klerk MT, Smeets PAM, la Fleur SE. Inhibitory control as a potential treatment target for obesity. Nutr Neurosci. 2023 May;26(5):429-444. doi: 10.1080/1028415X.2022.2053406. Epub 2022 Mar 28. PMID 35343884
- [Background] Keeler JL, Chami R, Cardi V, Hodsoll J, Bonin E, MacDonald P, Treasure J, Lawrence N. App-based food-specific inhibitory control training as an adjunct to treatment as usual in binge-type eating disorders: A feasibility trial. Appetite. 2022 Jan 1;168:105788. doi: 10.1016/j.appet.2021.105788. Epub 2021 Oct 30. PMID 34728250
- [Background] Cardi V, Meregalli V, Di Rosa E, Derrigo R, Faustini C, Keeler JL, Favaro A, Treasure J, Lawrence N. A community-based feasibility randomized controlled study to test food-specific inhibitory control training in people with disinhibited eating during COVID-19 in Italy. Eat Weight Disord. 2022 Oct;27(7):2745-2757. doi: 10.1007/s40519-022-01411-9. Epub 2022 Jun 6. PMID 35666376
- [Background] Bottesi G, Ghisi M, Altoe G, Conforti E, Melli G, Sica C. The Italian version of the Depression Anxiety Stress Scales-21: Factor structure and psychometric properties on community and clinical samples. Compr Psychiatry. 2015 Jul;60:170-81. doi: 10.1016/j.comppsych.2015.04.005. Epub 2015 Apr 15. PMID 25933937
- [Background] Calugi S, Milanese C, Sartirana M, El Ghoch M, Sartori F, Geccherle E, Coppini A, Franchini C, Dalle Grave R. The Eating Disorder Examination Questionnaire: reliability and validity of the Italian version. Eat Weight Disord. 2017 Sep;22(3):509-514. doi: 10.1007/s40519-016-0276-6. Epub 2016 Apr 2. PMID 27039107
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] Cepeda-Benito A, Gleaves DH, Fernandez MC, Vila J, Williams TL, Reynoso J. The development and validation of Spanish versions of the State and Trait Food Cravings Questionnaires. Behav Res Ther. 2000 Nov;38(11):1125-38. doi: 10.1016/s0005-7967(99)00141-2. PMID 11060941
- [Background] Stunkard AJ, Messick S. The three-factor eating questionnaire to measure dietary restraint, disinhibition and hunger. J Psychosom Res. 1985;29(1):71-83. doi: 10.1016/0022-3999(85)90010-8. PMID 3981480
- [Background] Gormally J, Black S, Daston S, Rardin D. The assessment of binge eating severity among obese persons. Addict Behav. 1982;7(1):47-55. doi: 10.1016/0306-4603(82)90024-7. PMID 7080884
- [Background] Innamorati M, Imperatori C, Manzoni GM, Lamis DA, Castelnuovo G, Tamburello A, Tamburello S, Fabbricatore M. Psychometric properties of the Italian Yale Food Addiction Scale in overweight and obese patients. Eat Weight Disord. 2015 Mar;20(1):119-27. doi: 10.1007/s40519-014-0142-3. Epub 2014 Jul 29. PMID 25069837
- [Background] Fossati A, Di Ceglie A, Acquarini E, Barratt ES. Psychometric properties of an Italian version of the Barratt Impulsiveness Scale-11 (BIS-11) in nonclinical subjects. J Clin Psychol. 2001 Jun;57(6):815-28. doi: 10.1002/jclp.1051. PMID 11344467
- [Background] Labonte K, Nielsen DE. Measuring food-related inhibition with go/no-go tasks: Critical considerations for experimental design. Appetite. 2023 Jun 1;185:106497. doi: 10.1016/j.appet.2023.106497. Epub 2023 Mar 7. PMID 36893916